CLINICAL TRIAL: NCT00904852
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation Study of Tandutinib (Formerly MLN518) in Combination With Temozolomide and Bevacizumab Following Concurrent Radiation Therapy and Temozolomide in the Treatment of Patients With Newly Diagnosed Glioblastoma Multiforme.
Brief Title: Safety Study of the Combination of Tandutinib With Temozolomide and Bevacizumab After Radiation and Temozolomide in Patients With Newly Diagnosed With Glioblastoma Multiforme
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Anthony Boral, Vice President Clinical Research, Millennium Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C03003
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — tandutinib; Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tandutinib, bevacizumab, and temozolomide (Experimental): tandutinib in combination with temozolomide and bevacizumab following concurrent radiation therapy and temozolomide treatment.
  Interventions: Drug: Tandutinib, bevacizumab, and temozolomide

INTERVENTIONS:
Drug: Tandutinib, bevacizumab, and temozolomide — All patients will have completed treatment with concurrent radiation therapy and temozolomide. Patients will be entered into different dosing groups of tandutinib. Patients will receive up to 6 cycles of treatment with oral temozolomide at 150 mg/m2 daily for the first 5 days of a 28 day cycle, oral tandutinib at escalating doses 250, 375, 500, or 625 mg twice daily on days 1 to 28, and intravenous bevacizumab at 10 mg/kg on days 1 and 15 of each cycle

SUMMARY:
This is a safety study of tandutinib in combination with temozolomide and bevacizumab after people have received radiation therapy and temozolomide treatment. This study will determine the maximum safe dose of tandutinib when combined with temozolomide and bevacizumab and evaluate the safety of the combination treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glioblastoma multiforme
* Received radiotherapy for glioblastoma multiforme
* Patients who have not had previous treatments for glioblastoma multiforme (except for surgery, radiation and temozolomide therapy)
* Females that are postmenopausal for at least 1 year prior to screening visit
* 18 years of age and older

Exclusion Criteria:

* Other brain cancers that are not diagnosed as glioblastoma multiforme
* female patients who are lactating or are pregnant
* HIV positive and/or any other active infection requiring therapy
* Known hepatitis B or hepatitis C infection
* Diagnosed or treated any other cancer within 2 years before the first dose
* History of cardiovascular conditions and/or vascular disease
* Allergic to any component of bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of tandutinib, adverse events, serious adverse events and dose limiting toxicities, clinical laboratory values and vital sign measurements | Cycle 1 days 1, 8, 15, and 22. Cycle 2 -6 days 1 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Parasuraman, MD, Study Director — Millennium Pharmaceuticals, Inc.